CLINICAL TRIAL: NCT02528838
Title: A Non-interventional Observational Post Authorization Study to Assess Safety and Outcome of the Various Medication Usage Patterns in Clinical Routine Practice in Patients Receiving Lenalidomide (REVIEW)
Brief Title: An Observational Study to Assess Safety and Outcome of the Various Medication Usage Patterns in Clinical Routine Practice in Patients Receiving Lenalidomide.
Acronym: REVIEW
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS-Celgene-NETH-001
Record Dates: First submitted 2015-08-06; First posted 2015-08-19 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Non-interventional; Observational; Lenalidomide; REVIEW; Post-authorization; Netherlands
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Revlimid according to clinical practice

SUMMARY:
The study is designed as a prospective, non-interventional, observational single arm study. Hundred-fifty patients over 18 with stable disease or at least partial response while on treatment with lenalidomide will be recruited from approximately 20 haematology/oncology sites in the Netherlands. Recruitment will continue until 150 patients have started the study. When this target is reached, all patients on lenalidomide will continue to be followed until the last patient has been followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who understand and voluntarily sign an informed consent form.
* Patients with multiple myeloma who are currently receiving lenalidomide treatment and who have taken lenalidomide for > 2 cycles and < 6 cycles.
* Patients with currently stable disease or meeting the criteria for complete response, very good partial response or partial response while on lenalidomide treatment.

Exclusion Criteria:

* Refusal to participate in the study.
* Women who are pregnant or breast-feeding.
* Women of childbearing potential unless all of the conditions of the Pregnancy Prevention Programme are met.
* Hypersensitivity to the active substance or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already successfully, i.e. with currently stable disease or meeting the criteria for complete response, very good partial response or partial response, on-treatment for maximally up to 6 cycles with lenalidomide at each site will be enrolled into the study. In all cases, the decision to treat the patient with lenalidomide was already made prior to the decision to enter the subject into the study.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) | Up to approximatly 4 years
  Adverse events will be classified using the MedDRA classification system. The severity of the toxicities will be graded according to the NCI CTCAE VERSION 4.03 whenever possible

SECONDARY OUTCOMES:
Quality of Life | Up to approximatly 24 months
  Quality of life will be measured by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire(EORTC QL Q-C30) and EORTC QLQ-MY20
Lenalidomide usage patterns | Up to approximatly 4 years
  Registration in case report form (CRF) and evaluation of usage patterns in daily clinical practice
Lenalodomide dose modifications | Up to approximatly 4 years
  Registration in case report form (CRF) and evaluation of dose modifications in daily clinical practice
Reasons for discontinuation of lenalidomide | Up to approximatly 4 years
  Registration in case report form (CRF) and evaluation of reasons of discontinuation in daily clinical practice
Clinical outcome | Up to approximately 4 years
  Clinical outcome will be measured using routine assessment criteria (i.e. IMWG)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Stevens, MSc, Study Director — Celgene BV